CLINICAL TRIAL: NCT06096974
Title: A Multi-Center, Open-Label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of Pan-RAS Inhibitor YL-17231 in Patients With Advanced Solid Tumors Harboring Mutations in KRAS, HRAS, or NRAS
Brief Title: Pan-RAS Inhibitor YL-17231 in Patients With Advanced Solid Tumors Harboring Mutations in KRAS, HRAS, or NRAS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YL-17231-001
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors
Keywords: KRAS, HRAS, or NRAS Mutations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): Dose escalation of YL-17231 to determine maximum tolerated dose.Expansion cohort to ensure sufficient safety experience, pharmacokinetic information, and early evidence of clinical activity of YL-17231 to recommend Phase 2 regimens
  Interventions: Drug: YL-17231

INTERVENTIONS:
Drug: YL-17231 — YL-17231 will be administered orally once daily in a continuous regimen

SUMMARY:
This study will evaluate the safety, tolerability, drug levels, pharmacodynamic effects, and clinical activity of YL 17231 in patients with advanced solid tumors harboring mutations in KRAS, HRAS, or NRAS.

DETAILED DESCRIPTION:
The study is a Phase 1, multi-center, open label study in 2 parts.

Part 1 (Phase Ia):

This is a 3 + 3 design dose escalation study, to evaluate the safety and tolerability, and to determine the MTD and/or RP2D of YL-17231 treatment when administered orally QD in patients with advanced solid tumors harboring mutations in KRAS, HRAS or NRAS. Up to 9 doses cohorts are planned for the dose escalation part of the study, with the starting dose of 0.25mg QD. The actual number of dose cohorts to be explored in this study will be determined by the non-tolerable dose based on dose limiting toxicities (DLTs) in conjunction with the PK and preliminary efficacy signal data. If suggested by safety and PK findings from planned dose treatment cohorts, additional dose levels may be evaluated and dosing interval may be modified under the Safety Monitoring Committee (SMC) guidance.

In Part 1, the 3+3 trial design for the dose escalation will be used and a total of 9 dose levels starting dose of 0.25 mg OD is planned.

One cycle is 21 days. DLT observation period is one cycle. The maximum tolerated dose (MTD) is the highest dose at which ≤1 of 6 patients experiences a DLT during the DLT observation period. The study will identify a maximum tolerated dose (MTD) if possible, with safety and tolerability data. All available data, including safety, tolerability, PK, PD and preliminary anti-tumor activity from each cohort will be reviewed by the SMC to determine the RP2D.

Patients may be permitted an intra-patient dose-escalation of YL-17231 to a higher dose level that has been cleared and deemed safe by the SMC if they have completed Cycle 2 at their initial enrolled dose level and continued on-study with no treatment related ≥ Grade 2 AEs. The Investigator must consult with the Medical Monitor to confirm if the patient is permitted be dose-escalated to a dose-level already cleared by the SMC.

Backfilling Additional patients (up to total of 12) may be enrolled in the dose levels which have been cleared and deemed safe by SMC to further evaluate the safety, tolerability and PK. This is referred to as backfilling.

Part 2 (Phase Ib):

This is a dose expansion phase to further evaluate the safety, tolerability and preliminary anti-tumor activity of YL 17231 at the RP2D selected by SMC.

The number of patients to be enrolled for the expansion cohorts, the RP2D and the desired patient population will be determined by the emerging data from part 1 of the study, including safety, tolerability, PK, PD and preliminary anti-tumor efficacy, as well as any other relevant evolving clinical data, and will be clarified through a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic advanced solid tumors with no standard therapies, or having progressed on or intolerable to standard therapies.
* Advanced solid tumors harboring mutations in KRAS, HRAS or NRAS as determined by laboratory testing, including local laboratory testing.
* Measurable disease with at least one lesion amenable to response assessment per RECIST 1.1.
* Demonstrate adequate organ function as defined below. All screening laboratories should be performed within 7 days of study treatment initiation.

  1）Absolute neutrophil count (ANC) ≥1.2 × 10^9/L；2）Platelets ≥100 × 10^9/L Hemoglobin ≥9 g/dL or ≥5.6 mmol/L；3）Measured or calculated creatinine clearance (CrCl)(Cockcroft-Gault) ≥60 mL/min；4）Total bilirubin ≤1.5 × ULN (patients with Gilbert's syndrome, total bilirubin ≤3.0 × ULN) ；5）Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN or ≤5 × ULN for patients with liver metastases
* Has an ECOG performance status of 0-1.
* Life expectancy ≥12 weeks at baseline.
* Women of childbearing potential must have negative serum or urine pregnancy test within 72 hours prior to receiving the first study drug administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* For women of childbearing potential, must be willing to use an adequate method of contraception from 30 days prior to the first study drug administration and at least 3 months following last day study drug administration.
* Male patients of childbearing potential must be surgically sterile, or must agree to use adequate method of contraception during the study and at least 3 months following the last day of study drug administration.
* Age ≥18 years at screening.
* Able and willing to provide written informed consent and to follow study instructions.
* Washout from prior anti-tumor therapy:1）Cytotoxic therapies ≥ 3 weeks Mitomycin C or nitrosoureas ≥ 6 weeks；2）Small molecule agents ≥2 weeks or 5x T1/2, whichever is longer；3）Biologic agents (e.g., antibodies) ≥ 4weeks Immunotherapy (e.g., CTLA4, PD-1, PD-L1 inhibitors) ≥ 4 weeks；4）Radiotherapy ≥ 4 weeks；5）Limited field radiotherapy or palliative radiotherapy ≥ 2 weeks ；6）Major surgery, excluding biopsy ≥ 4 weeks (exception: patients may enroll if fully recovered or without intolerable or clinically significant adverse effects, but at least 14 days must have elapsed between major surgery and first study drug administration)；7）Study drug with an investigational product, or non-approved use of a drug or device ≥ 4 weeks (≥2 weeks or 5x T1/2, whichever is longer for small molecule agents

Exclusion Criteria:

* Known symptomatic brain metastases requiring dexamethasone ≥4mg (or equivalent) or requiring steroid dose increase within 14 days prior to the first dose of YL-17231.
* Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment.
* Unresolved toxicities from prior therapy, defined as having not resolved to NCI CTCAE v.5.0 Grade ≤1 1 or baseline, with exception of endocrinopathies from prior therapy and successfully treated (such as hypothyroidism), alopecia, vitiligo, and ≤ grade 2 peripheral neuropathy.
* Human immunodeficiency virus (HIV) infection with a current or a known history of AIDS-defining illness or HIV infection with a CD4+ T cell count <350 cells/µL and an HIV viral load more than 400 copies/µL.
* Patients with active viral (any etiology) hepatitis are excluded. However, patients with serologic evidence of chronic hepatitis B virus (HBV) infection (defined by a positive hepatitis B surface antigen test and a positive anti-hepatitis core antigen antibody test) who have a viral load below the limit quantification (HBV DNA titer <1000 cps/mL or 200 IU/mL), and are not currently on viral suppressive therapy may be eligible and should be discussed with the Medical Monitor. Patients with a history of hepatitis C virus (HCV) infection who have completed curative antiviral treatment and have a viral load below the limit of quantitation may be eligible and should be discussed with the Medical Monitor.
* Any of the following cardiac criteria experienced currently or within the last 6 months:

  1. Congestive heart failure (New York Heart Association ≥ Class 2).
  2. Any clinically significant abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting electrocardiograms (ECGs), e.g., complete left bundle branch block or third-degree heart block.
  3. Acute coronary syndrome within 6 months.
  4. Clinically significant cardiac arrhythmia.
* Mean QTC interval corrected (Frederica) for heart rate >450 ms.
* Left ventricular ejection fraction (LVEF) <50% or the lower limit of normal (per institutional standard).
* Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection, as determined by the investigator.
* Any condition that impairs a patient's ability to swallow whole pills. Presence of an active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of YL-17231, as determined by the investigator.
* History noninfectious pneumonitis required steroids treatment or concurrent pneumonitis or interstitial lung diseases.
* An active additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Known allergy to any component of YL-17231.
* Patient has known psychiatric, substance abuse or other disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the investigator.
* Patients who are pregnant or breastfeeding or expecting to conceive within the projected duration of the trial, starting with the screening visit through 3 months after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities (DLTs) | The first cycle (21 days)
  A toxicity will be considered dose-limiting if it occurs during the first cycle (21 days) of treatment with YL-17231.
TEAEs | Through study completion, an average of 1 year
  AEs will be coded using Medical Dictionary for Regulatory Activities current version. AEs will be regarded as treatment-emergent AEs (TEAEs) if they occur after first treatment. The frequencies will be presented including number and percentages of patients having experienced an event and the total number of events.
SAEs | Through study completion, an average of 1 year
  Serious AEs

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From first dose of study treatment to the first documented disease progression or death due to any cause, whichever occurs first， assessed up to 30 months.
  ORR, defined as percentage of patients with a documented CR or PR in Response Evaluation Criteria in Solid Tumors 1.1(RECIST 1.1)
Duration of Response (DOR) | From first documentation of a response (PR or CR) to the first documented disease progression or death due to any cause, whichever occurs first， assessed up to 30 months.
  DOR, defined as time from first documentation of a response (PR or CR) to the first documented disease progression or death due to any cause, whichever occurs first, for those patients with a PR or CR.
Progression Free Survival (PFS) | From first dose of study treatment to the first documented disease progression or death due to any cause, whichever occurs first, assessed up to 30 months.
  PFS, defined as time from first dose of study treatment to the first documented disease progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | From first dose of study treatment to the first documented disease progression or death due to any cause, whichever occurs first, assessed up to 30 months.
  DCR, defined as percentage of patients with a documented CR or PR and SD
AUC(0-T) | During Cycles 1 and 2 (each cycle is 21 days)
  Area under the concentration-time curve from time zero to the last quantifiable concentration of YL-17231
Cmax | During Cycles 1 and 2 (each cycle is 21 days)
  Maximum observed serum concentration of YL-17231 is observed directly from data
T1/2 | During Cycles 1 and 2 (each cycle is 21 days)
  Elimination half life of YL-17231 is observed directly from data
Tmax | During Cycles 1 and 2 (each cycle is 21 days)
  Time to maximum plasma concentration of YL-17231 is observed directly from data as time of Cmax

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute and Hospital, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No